CLINICAL TRIAL: NCT07159711
Title: Evaluation of Seismocardiography (SCG) as a Tool for Assessing Fitness and Predicting Outcomes in Oesophageal Cancer Surgery
Brief Title: Evaluation of Seismocardiography(SCG) for Assessing Fitness and Predicting Outcomes in Oesophageal Cancer Surgery
Acronym: SEISMIC
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 342434
Record Dates: First submitted 2025-07-17; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Oesophageal Cancer; Oesophageal Adenocarcinoma; Prehabilitation; Oesophagectomy; Neoadjuvant Chemotherapy
Keywords: oesophageal cancer; Oesophagectomy; Fitness; Prehabilitation; Neoadjuvant chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Seismofit — Seismofit® is a 3 x 5 x 1.5 cm Class I medical device manufactured by Ventriject, which utilizes SCG principles and machine learning to estimate an individual's fitness. It is afixed to a patient's sternum with an adhesive patch. It measures the amplitude and timing of vibrations on the chest using accelerometers. The device then averages the data collected over 45 seconds to create the SCG. From the SCG, several maxima and minima (fiducial points) are identified, which correlate to the opening and closing of the mitral and aortic valves. Features of the SCG, including the timing, frequency, amplitude, and variability of these points, are then incorporated into an algorithm that also considers patient height, weight, age, and sex to calculate the VO2 peak.
  Data is transmitted via Bluetooth to an allocated smartphone app.
  Other Names: Seismocardiography based VO2 Max Estimation of Fitness

SUMMARY:
Oesophageal cancer is a common cause of cancer death worldwide. Curative treatment involves chemotherapy and surgery but has significant risks. Therefore, patient selection and improving physical fitness to withstand such major treatment is important to reduce the risk of complications. Physical fitness is traditionally measured by a specialised exercise test called Cardiopulmonary exercise testing (CPET), which can take up to one hour and requires specialised staff and expensive equipment such as a graded exercise bike or treadmill. Seismofit is a small device (smaller than a smartphone) used to estimate fitness in patients in under three minutes while lying down at rest. It measures the vibrations generated by the heart and, together with patient height, weight, age, and gender, accurately estimates fitness using an algorithm developed in healthy patients. The device has never been tested in a large group of oesophageal cancer patients to see if it can be used to predict complications in patients undergoing cancer treatment.

In this study, patients undergoing Oesophageal cancer treatment with chemotherapy or chemoradiotherapy and surgery will have Seismofit measurements at various points during their treatment to see if we can predict complications and hospital stay. Secondly, this study will also evaluate the accuracy of Seismofit compared to the gold standard CPET results in cancer patients.

DETAILED DESCRIPTION:
Oesophageal cancer is the 8th most common cause of cancer and the 6th leading cause of cancer-related deaths worldwide(West et al., 2016; Liu et al., 2023). Surgery with curative intent has been associated with significant morbidity and mortality despite recent advancements in anaesthesia and surgical techniques(Wu et al., 2014). Good patient selection with optimisation of cardiorespiratory fitness (CRF) is essential to improve surgical outcomes(West et al., 2014; Ozova et al., 2022). This is particularly important given that most oesophageal cancer patients undergo neo-adjuvant treatment (e.g. chemotherapy), which is known to have a significant adverse effect on patient fitness before surgery (mean reduction of 12.1% in VO2Peak) (Jack et al., 2014). A lower baseline level of fitness has also been shown to be associated with morbidity and mortality in patients undergoing treatment with curative intent (Hennis et al., 2011; West et al., 2024). Prehabilitation is now considered the standard of care in oesophageal cancer surgery, with societal guidance recently recommending a baseline fitness assessment to tailor the intervention as well as a means of monitoring response (Walker et al., 2024).

Cardiopulmonary Exercise Testing (CPET) is considered the gold standard in measuring the CRF of an individual by obtaining the maximal volume of oxygen consumed (VO2Peak) in samples of expired gas during a graded effort cycle ergometer test (Krogh et al., 2020; Levett et al., 2018a). However, CPET is a resource-intensive, costly, time-consuming test (requiring up to 60 minutes) and creates a significant time burden on patients with already busy treatment schedules. In a UK survey of prehabilitation practice, 50% of Upper Gastrointestinal (UGI) units used CPET at baseline, with only 80% of these (40% total) using CPET for response assessment (Barman et al. 2024 in revision for publication Annals RCS Eng).

Seismofit® is a device that accurately estimates the VO2Peak using machine learning algorithms incorporating seismocardiography (SCG) and patient parameters such as height, weight, age, and gender. SCG is a process by which vibrations generated by the heart during its regular physiological cycles are characterised and mapped for changes in morphology, frequency, intensity and character(Sørensen et al., 2018). Key advantages of Seismofit® include its inter-test reliability, rapid availability of results (i.e., estimation of fitness in under 3 minutes in an outpatient setting), and accurate estimation of fitness in a resting patient (Hansen et al., 2023a). The accuracy of Seismofit® in comparison to CPET-measured CRF has previously been demonstrated with a Mean Absolute Percentage Error (MAPE) of 12.3% in healthy adult populations(Hansen et al., 2023b). However, there is minimal data on cancer patients, and no studies have correlated VO2Peak generated by Seismofit® to clinical outcomes.

Given the potential benefits of Seismofit® over CPET, this study will investigate its validity in a clinical setting across four major Oesophageal cancer resection centres (Guy's and St Thomas NHS Foundation Trust (GSTT), University Hospitals Southampton (UHS), Royal Marsden NHS Foundation Trust (RM) and Royal Surrey NHS Foundation Trust (RS).

This will be the first study to evaluate the use of Seismofit® in a large volume of oesophageal cancer patients. With correlation to clinical outcomes, this study will serve as the basis for future research into the use of Seismofit® in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* Diagnosis of Oesophageal cancer (T0-4 N0-3 M0, Oesophageal / Gastro-Oesophageal Junction (GOJ) type 1-2 adenocarcinoma
* Patients being considered for curative treatment (i.e. due to undergo NAC and Oesophagectomy / Oesophago-Gastrectomy [open / MIO / hybrid / robotic])
* Patients able to give informed consent

Exclusion Criteria:

* Pregnant patients.
* Patients under the age of 18.
* Patients undergoing primary Oesophagectomy +/- Oesophago-Gastrectomy with no neoadjuvant therapy.
* Patients undergoing Neoadjuvant chemoradiotherapy.
* Patient's being treated with curative intent for Oesophageal Squamous cell carcinoma
* Patients that are deemed not fit or suitable for Oesophagogastric cancer resection as part of a Multi-Disciplinary Team meeting decision.
* Patients with implanted devices such as pacemakers or cardioverter-defibrillators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be patients undergoing treatment for oesophageal cancer with curative intent that meet the above outlined inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of pneumonia as defined by the Esophageal Complications Consensus Group criteria (ECCG). | 2 Years
  This study will evaluate whether fitness and changes in the Seismofit estimated VO2Max through the treatment period will be able to predict increased rates of pneumonia.
Overall rate of complications as defined by the Clavien-Dindo classification | 2 Years
  This study will evaluate whether fitness and changes in the Seismofit estimated VO2Max through the treatment period will be able to predict increased overall complications as well overall major complications defined as Clavien-Dindo Classification of III and above.
Total hospital length of stay for patients being treated for Oesophageal cancer | 2 Years
  This study will evaluate whether fitness and changes in the Seismofit estimated VO2Max will be able to predict increased hospital length of stay.

SECONDARY OUTCOMES:
Seismofit® estimated VO2Peak reading accuracy compared to "gold standard" CPET measured VO2Peak. | 2 Years
  This study will evaluate the association between Seismofit® estimated VO2Peak to the gold standard CPET measured VO2Peak.
To compare if Seismofit® is able to stratify patients into the lower quartiles of fitness accurately based on CPET measured fitness. | 2 Years
  This study will evaluate whether Seismofit® is able to accurately stratify patients into the same quartiles of fitness as CPET.
To investigate Seismofit® estimated fitness and Chemotherapy compliance & tolerability. | 2 Years
  This study will investigate whether patients with higher Seismofit estimated VO2Max will tolerate neoadjuvant chemotherapy better than those classified within the lower levels of fitness.
ITU length of stay (and re-admission) | 2 Years
  This study will investigate whether patients with lower Seismofit estimated VO2Max, and more rapid decline in this fitness after Oesophagectomy will have longer lengths of stay in Intensive Treatment Units (ITU) or have higher return to ITU when they are stepped down to ward level care.
Anastomotic leak rates | 2 Years
  This study will investigate whether patients with lower Seismofit estimated VO2Max, and more rapid decline in this fitness after Oesophagectomy will have higher anastomotic leak rates.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD FRCS, Principal Investigator — Guy's and St Thomas NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
All collected pseudonymised datapoints that underlie results in publication will be shared. The individual consent forms will be stored at each of the research sites. At the time of upload to the REDCap research database, a case reporting form code number will be generated. Patient identifiable information will not leave the research site at which the patient receives treatment.
Supporting Information: SAP, ICF, CSR
Time Frame: June 2025
Access Criteria: Only local research teams will have access to patient-identifiable data. The central research team at GSTT will have access to pseudonymized data, except for patients recruited locally at GSTT. At the time of upload onto REDCap by the local research team, a case number will be used to pseudonymise patient data. This case number will be recorded on the consent form and may be used if research teams need to trace and link back to the patient.
  Consent forms will be stored in a secure NHS computer system folder at each local research site or, where paper forms are used, in a secure locker. In the event paper case reporting forms are used, they will also be stored similarly to the paper consent forms in a secure locker. In both electronic and physical cases, access to patient-identifiable documentation will be limited to the local PI/trial manager and other authorised personnel (research students, nursing staff, etc.) involved in the data set's collection, verification or analysis.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT07159711/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT07159711/ICF_001.pdf